CLINICAL TRIAL: NCT07370714
Title: A Multicenter, Prospective, Observational Study on Factors Affecting Wound Dehiscence in Pilonidal Sinus Surgery: The Impact of Anal Proximity, Morphological Stage, and Surgical Technique (ORIPIS)
Brief Title: Factors Affecting Wound Dehiscence in Pilonidal Sinus Surgery (ORIPIS)
Status: Recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Bahattin Bayar, Specialist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK-2025-290
Record Dates: First submitted 2025-12-23; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pilonidal Sinus Disorder
Keywords: pilonidal sinus; risk factors; surgical wound dehiscence; Surgical Closure Technique
MeSH Terms: conditions — Pilonidal Sinus; Surgical Wound Dehiscence | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months

GROUPS / COHORTS (1):
- Pilonidal Sinus Surgery Patients: This cohort includes adult patients undergoing pilonidal sinus surgery as part of routine clinical care at participating centers. The study is observational in nature, and no experimental intervention is assigned. Surgical technique, anatomical characteristics including proximity to the anal verge, and morphological stage of the disease are determined by the treating surgeon according to standard practice. Patients are prospectively followed after surgery, and postoperative wound outcomes are recorded for observational analysis.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — This is an observational study. No experimental intervention is assigned. Surgical procedures are performed as part of routine clinical care according to standard practice and are not determined by the study protocol.

SUMMARY:
The goal of this multicenter, prospective, observational study is to investigate factors associated with wound dehiscence following pilonidal sinus surgery. The main questions it aims to answer are:

Does the proximity of the pilonidal sinus to the anal verge influence the risk of postoperative wound dehiscence? How do the morphological stage of the disease and the surgical technique used affect wound healing outcomes? Patients undergoing pilonidal sinus surgery as part of routine clinical care will be enrolled prospectively across multiple centers. Clinical, anatomical, and surgical characteristics-including anal proximity, morphological stage, and type of surgical technique-will be recorded. Participants will be followed postoperatively, and wound outcomes will be assessed to identify factors associated with wound dehiscence.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age)
* Diagnosis of pilonidal sinus disease
* Patients undergoing pilonidal sinus surgery as part of routine clinical care
* Ability to provide informed consent

Exclusion Criteria:

* Patients undergoing emergency surgery
* Previous pilonidal sinus surgery at the same site
* Inability to complete postoperative follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with pilonidal sinus disease who undergo pilonidal sinus surgery as part of routine clinical care at participating centers. Eligible patients are enrolled prospectively and followed after surgery. Demographic, anatomical, and surgical characteristics are recorded for observational analysis of postoperative wound outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Wound Dehiscence | Within 30 days after surgery
  Wound dehiscence is defined as partial or complete separation of the surgical wound occurring after pilonidal sinus surgery, as assessed during postoperative follow-up.

SECONDARY OUTCOMES:
Time to Complete Wound Healing | Up to 90 days after surgery
  Time from surgery to complete epithelialization of the surgical wound without discharge or need for additional intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made publicly available. De-identified data may be shared for scientific purposes upon reasonable request, in accordance with institutional policies and ethics committee approval.